CLINICAL TRIAL: NCT06208397
Title: Noninvasive Evaluation in Diagnosis and Treatment of Histopathological Growth Patterns in Colorectal Liver Metastases Using MR Elastography-based Shear Strain Mapping
Brief Title: MRE for Assessment of Histopathological Growth Patterns in Colorectal Liver Metastases
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yu Shi, Deputy director of department of radiology, Shengjing Hospital
Other Study IDs: ShengjingH-CRLM2023
Record Dates: First submitted 2024-01-06; First posted 2024-01-17 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer liver metastasis; Magnetic Resonance Imaging; Magnetic Resonance Elastography; Histopathological growth patterns
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Diagnostic (MRE): Patients undergo a preoperative routine MRI scan and MRE the day before their scheduled surgery to assess OSS and NOSS. After surgery, the HGP of tumor will be assessed by H&E-stained sections.
  Interventions: Diagnostic Test: Magnetic Resonance Elastography and routine MRI

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Elastography and routine MRI — Assessed boundary conditions through MRE-base SII before surgery and recorded HGP of tumor after surgery.
  Other Names: MRE

SUMMARY:
The goal of this study is to investigate the value of MR elastography-based SII as a means of detecting HGP noninvasively in patients with pathology-proven CRLM. MRE will provide a direct measure of tumor-liver adhesion to investigate the relationship between imaging findings and pathophysiological changes in the Liver.

DETAILED DESCRIPTION:
Colorectal cancer ranks third in terms of incidence and second in terms of mortality among all cancers on the global cancer burden, based on the GLOBOCAN 2020 estimates. Among people diagnosed with colorectal cancer, 20% have metastatis, and 40% present with recurrence after previously treated localized disease. Liver is the most common site of metastasis besides lymph nodes, with a 5-year survival rate of less than 20%. Histopathological growth patterns (HGPs) appear at the interface between the tumour border and surrounding liver parenchyma which can be identified by light microscopy on tissue sections. Three primary HGPs have been identified: desmoplastic HGP (dHGP), replacement HGP and the pushing HGP. In the dHGP, the cancer cells are separated from the liver by a capsule of desmoplastic stroma in which new blood vessels are formed by sprouting angiogenesis. Recently, it has been reported that dHGP is linked to a better outcome in terms of survival and more clinical benefit achieved with preoperative anti-angiogenic therapy in patients with colorectal cancer liver metastasis (CRLM). Thus, planning of preoperative treatment might greatly benefit from HGP prediction. Preoperative prediction of HGP is challenging, however, as HGP is a histopathologic finding that can be diagnosed only with a postoperative surgical specimen. Previous studies have made many efforts to identify HGP through radiologic features (e.g., tumor margin, perilesional rim enhancement, or fused radiomics signature) by CT or MRI. However, high variability was observed in the assessment of these imaging characteristics, and they did not provide a direct measure of tumor-liver adhesion, leading to controversy in clinical practice. Recently, an MRE-based technique, termed "slip interface imaging" (SII), has been used to quantify the degree of tumor-peritumoral tissue adhesion in brain tumors and microvascular invasion in hepatocellular carcinoma noninvasively, may have the potential to characterize the mechanical characteristics of the tumor-liver interface and predict HGP of CRLM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed CRLM
* Pathologic results obtained in surgical patients
* No contraindications for magnetic resonance imaging examination

Exclusion Criteria:

* Image quality does not meet the measurement requirements.
* the diameter of CRLM <1cm
* Combined with other important organ dysfunction
* Combined with malignant tumor
* Patients who do not sign an informed consent
* Patients with metallic implants or foreign bodies in their bodies (pacemakers, artificial metallic heart valves, metal joints, metal implants, and those who cannot remove dentures, insulin pumps, or contraceptive rings)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subject inclusion criteria were adult patients with CRLM.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-24 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Radiological assessment of CRLM | Baseline to 6 weeks
  Examinations were performed on a 3.0T MRI. Mechanical vibration frequencies of 30 and 60 Hz were applied in synchrony with the MRE pulse sequence. Regions of interest (ROIs) were placed manually in the liver. The performance of the use of SII to predict HGP of tumor was evaluated with the Wilcoxon rank sum, 1-way ANOVA, and Tukey-Kramer tests.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Shi, M.D., Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Latacz E, Hoppener D, Bohlok A, Leduc S, Tabaries S, Fernandez Moro C, Lugassy C, Nystrom H, Bozoky B, Floris G, Geyer N, Brodt P, Llado L, Van Mileghem L, De Schepper M, Majeed AW, Lazaris A, Dirix P, Zhang Q, Petrillo SK, Vankerckhove S, Joye I, Meyer Y, Gregorieff A, Roig NR, Vidal-Vanaclocha F, Denis L, Oliveira RC, Metrakos P, Grunhagen DJ, Nagtegaal ID, Mollevi DG, Jarnagin WR, D'Angelica MI, Reynolds AR, Doukas M, Desmedt C, Dirix L, Donckier V, Siegel PM, Barnhill R, Gerling M, Verhoef C, Vermeulen PB. Histopathological growth patterns of liver metastasis: updated consensus guidelines for pattern scoring, perspectives and recent mechanistic insights. Br J Cancer. 2022 Oct;127(6):988-1013. doi: 10.1038/s41416-022-01859-7. Epub 2022 Jun 1. PMID 35650276
- [Background] Frentzas S, Simoneau E, Bridgeman VL, Vermeulen PB, Foo S, Kostaras E, Nathan M, Wotherspoon A, Gao ZH, Shi Y, Van den Eynden G, Daley F, Peckitt C, Tan X, Salman A, Lazaris A, Gazinska P, Berg TJ, Eltahir Z, Ritsma L, Van Rheenen J, Khashper A, Brown G, Nystrom H, Sund M, Van Laere S, Loyer E, Dirix L, Cunningham D, Metrakos P, Reynolds AR. Vessel co-option mediates resistance to anti-angiogenic therapy in liver metastases. Nat Med. 2016 Nov;22(11):1294-1302. doi: 10.1038/nm.4197. Epub 2016 Oct 17. PMID 27748747
- [Background] Li M, Yin Z, Hu B, Guo N, Zhang L, Zhang L, Zhu J, Chen W, Yin M, Chen J, Ehman RL, Wang J. MR Elastography-Based Shear Strain Mapping for Assessment of Microvascular Invasion in Hepatocellular Carcinoma. Eur Radiol. 2022 Jul;32(7):5024-5032. doi: 10.1007/s00330-022-08578-w. Epub 2022 Feb 11. PMID 35147777
- [Background] Yin Z, Lu X, Cohen Cohen S, Sui Y, Manduca A, Van Gompel JJ, Ehman RL, Huston J 3rd. A new method for quantification and 3D visualization of brain tumor adhesion using slip interface imaging in patients with meningiomas. Eur Radiol. 2021 Aug;31(8):5554-5564. doi: 10.1007/s00330-021-07918-6. Epub 2021 Apr 14. PMID 33852045